CLINICAL TRIAL: NCT01054690
Title: A Comparative Study to Investigate if Silver Alloyed Urinary Catheters Can Reduce the Incidence of Catheter Acquired Urinary Tract Infections in Patients Undergoing Elective Surgery
Brief Title: Silver Alloyed Urinary Catheters and Incidence of Catheter Acquired Urinary Tract Infections (UTI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Bactiguard AB, Sweden (Unknown)
Responsible Party: Karin Stenzelius, PhD Nurse, Department of Urology, University Hospital in Lund
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H15 315/2007
Record Dates: First submitted 2010-01-14; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Urinary Tract Infection
Keywords: Catheterization; Urinary Tract Infection; Elective Surgery
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver alloyed urinary catheter (Experimental)
  Interventions: Device: Bactiguard Infection Protection (BIP) Cathter.
- Silicone urinary catheter (Placebo Comparator)
  Interventions: Device: Silicone Urinary Catheter

INTERVENTIONS:
Device: Bactiguard Infection Protection (BIP) Cathter.
  Arms: Silver alloyed urinary catheter
Device: Silicone Urinary Catheter
  Arms: Silicone urinary catheter

SUMMARY:
This study is a single blinded (Outcome Assessors), multicenter randomized controlled study designed to investigate if a silver alloyed urinary catheter with antibacterial properties can reduce the incidence of catheter acquired urinary tract infections in patients undergoing elective surgery. Patients requiring urinary catheterization will be randomized into two groups and receive either the silver alloyed catheter (test) or a silicone catheter (control).

ELIGIBILITY:
Inclusion Criteria:

* Adults in elective surgery requiring urinary catheterization

Exclusion Criteria:

* Patients who has or recently (within 3 weeks) had a urinary catheter
* Signs of urinary tracts infection
* Previous radiation therapy in lower pelvis
* Latex allergy
* Cognitive impaired
* Do not understand Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To determine whether a silver alloyed catheter with antibacterial properties will decrease the incidence of catheter associated urinary tract infection in patients undergoing elective surgery. | At catheter withdrawal (normally 1-3 days after catheter insertion).

SECONDARY OUTCOMES:
Patient´s evaluation of the catheterization and overall satisfaction. | At catheter withdrawal and 7-10 days after catheter withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Stenzelius, PhD Nurse, Principal Investigator — Department Urology, University Hospital in Lund, Sweden
Locations (3):
- Sweden (3):
  - Ortopedkliniken, Hässleholms Sjukhus, Hässleholm
  - Ortopedklinien, Lunds Hospital, Lund
  - Ortopedkliniken Lasarettet i Trelleborg, Trelleborg